CLINICAL TRIAL: NCT07208812
Title: Impact of Impression Techniques on Patient Satisfaction and Chewing Efficiency in 3D-Printed Implant Overdentures: A Crossover Study
Brief Title: 3D-Printed Implant Overdentures: Comparing Impression Techniques
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Shimaa Ebrahim Abo Elenin Ebrahim, Clinical demonstrator at prosthodontics department, Mansoura University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS.25.05.25
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-09

CONDITIONS: Edentulism
Keywords: 3D-Printed Implant Overdenture; Impression Techniques; Chewing Efficiency; Patient Satisfaction
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- conventional open -tray impression (Experimental): Mandibular implant overdenture fabricated using the conventional open tray impression technique at the implant level.
  Interventions: Procedure: Conventional open -tray impression
- Functionally generated reline impression (Experimental): Mandibular implant overdenture fabricated using functionally generated reline impression technique.
  Interventions: Procedure: Functionally generated reline impression
- Mucostatic base with functional borders impression (Experimental): Mandibular implant overdenture fabricated using mucostatic base and functional borders impression technique.
  Interventions: Procedure: Mucostatic base with functional borders impression

INTERVENTIONS:
Procedure: Conventional open -tray impression — Primary impression with irreversible hydrocolloid, custom tray with open window, and final impression with silicone material around impression copings to fabricate a 3D-printed implant overdenture
  Arms: conventional open -tray impression
Procedure: Functionally generated reline impression — Interim prosthesis relieved and reline impression taken during centric closure with border molding, scanned to construct a 3D-printed implant overdenture
  Arms: Functionally generated reline impression
Procedure: Mucostatic base with functional borders impression — Intraoral scan of edentulous arch, 3D-printed baseplates for occlusion rim, functional border molding, and digital workflow to fabricate 3D-printed implant overdenture
  Arms: Mucostatic base with functional borders impression

SUMMARY:
This randomized crossover clinical trial aims to compare three different impression techniques for the construction of 3d-printed mandibular implant overdentures in completely edentulous patients. Sixteen patients will receive two mandibular implants and three overdentures fabricated using:(1) conventional open-tray implant level impression (2) functionally generated reline impression, and (3)mucostatic base with functional borders impression. Each overdenture will be worn for three months with a washout period between interventions.

The primary outcome is masticatory efficiency, assessed using a color -mixing ability test at 3,6, and9 months.

Secondary outcome is patient satisfaction, assessed using a Visual Analog Scale (VAS) at the same intervals. the study hypothesis is that the impression technique influences both chewing efficiency and patient satisfaction

DETAILED DESCRIPTION:
Edentulism has a significant impact on oral function and quality of life. The use of mandibular implant overdentures supported by two implants is widely considered the minimum standard of care, providing improved stability, function, and patient satisfaction compared with conventional complete dentures. Recently, digital workflows and additive manufacturing (3D printing) have created new opportunities for fabricating complete dentures with improved efficiency and reduced costs.

Several impression techniques are currently available for implant-retained overdentures, but there is limited evidence on how these techniques influence functional outcomes and patient-reported satisfaction, particularly when using 3D-printed prostheses.

This randomized crossover clinical trial will be conducted at the Faculty of Dentistry, Mansoura University. Sixteen completely edentulous patients aged 45-70 years will receive two implants placed in the mandibular canine region. After the osseointegration period, each participant will be provided with three different mandibular implant overdentures fabricated using different impression techniques:

1. Conventional open-tray implant-level impression
2. Functionally generated reline impression
3. Mucostatic base with functional borders impression Each overdenture will be worn for a period of three months, with a two-week washout period using a provisional denture before switching to the next overdenture. Randomization will determine the sequence of interventions for each patient.

The primary outcome is masticatory efficiency, measured with a color-mixing ability test at 3, 6, and 9 months. The secondary outcome is patient satisfaction, measured using a Visual Analog Scale (VAS) at the same intervals.

The study is designed to provide evidence on whether the choice of impression technique affects clinical and patient-centered outcomes in 3D-printed mandibular implant overdentures.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients, free from systemic diseases that affect bone resorption (e.g., uncontrolled diabetes, osteoporosis)
* Residual alveolar ridges covered with healthy, firm mucosa
* Adequate mandibular bone length and width to accommodate standard implant sizes.
* Angle's Class I maxillo-mandibular relationship.

Exclusion Criteria:

* Absolute contraindications to implant placement (e.g., active cancer, immune system diseases)
* History of head and neck irradiation or chemotherapy within the past 3 years
* Metabolic bone diseases such as uncontrolled diabetes, osteoporosis, or hyperparathyroidism
* Parafunctional habits such as bruxism or clenching
* Smoking or alcoholism
* Any physical or medical condition that may interfere with study follow-up or implant success

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-01-06 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Masticatory efficiency | 3, 6, and 9 months after overdenture insertion
  Assessment of chewing efficiency using a color- mixing ability test

SECONDARY OUTCOMES:
Patient satisfaction | 3, 6, and 9 months after overdenture insertion
  Patient- reported satisfaction measured using the Visual Analog Scale

CONTACTS AND LOCATIONS:
Overall Officials: Shimaa E Aboelenin, Principal Investigator — Faculty of Dentistry, Mansoura University
Locations (1):
- Faculty of Dentistry, Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No